CLINICAL TRIAL: NCT05990192
Title: SOPRANO: Stereotactic Radiotherapy Alone or Followed by Niraparib for Oligometastases or Oligoprogression in Ovarian Cancer Following PARP Inhibitor Therapy
Brief Title: SBRT Alone or Followed by Niraparib for Oligometastases or Oligoprogression in Ovarian Cancer Following PARPi Therapy
Acronym: SOPRANO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICR-CTSU/2022/10082; 2022-003175-42 (EudraCT Number); CCR5726 (Other: RM/ICR Committee for Clinical Research); 23/LO/0719 (Other: London - Brighton & Sussex Research Ethics Committee)
Record Dates: First submitted 2023-06-21; First posted 2023-08-14 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Ovarian Cancer Recurrent
Keywords: Ovarian Cancer; Oligoprogressive; Oligometastatic; SBRT; PARP Inhibitor
MeSH Terms: conditions — Ovarian Neoplasms | interventions — niraparib; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SBRT followed by Niraparib (Other): SBRT treatment will commence within 7 days post randomisation and will be administered as detailed in the SOPRANO Radiotherapy Planning and Delivery Guidelines document. Doses will vary between 3 fractions over 5 days to 8 fractions over 19 days depending on the location of the lesions being treated.
  Niraparib treatment will start 4 weeks post completion of SBRT treatment and will continue daily until disease progression or other discontinuation criteria are met. Niraparib comes in oral tablet form and the starting dose will be 200mg per day (once a day) or 300mg per day (once a day) calculated by participant's weight and platelet count.
  Interventions: Drug: Niraparib oral capsule; Radiation: SBRT
- SBRT alone (Other): SBRT treatment will commence within 7 days post randomisation and will be administered as detailed in the SOPRANO Radiotherapy Planning and Delivery Guidelines document. Doses will vary between 3 fractions over 5 days to 8 fractions over 19 days depending on the location of the lesions being treated.
  Interventions: Radiation: SBRT

INTERVENTIONS:
Drug: Niraparib oral capsule — Niraparib used following SBRT treatment until disease progression
  Other Names: Zejula
  Arms: SBRT followed by Niraparib
Radiation: SBRT — SBRT may be delivered using a specialist SBRT platform, such as CyberKnife or with a linear accelerator with SBRT capabilities.
  Other Names: Stereotactic Body Radiotherapy

SUMMARY:
SOPRANO is a multi-centre, randomised phase II trial which aims to assess the impact of Stereotactic radiotherapy (SBRT) and continuing treatment with a PARP inhibitor (PARPi) for patients with oligometastatic or oligoprogressive ovarian, fallopian tube and primary peritoneal carcinoma. SOPRANO will also establish the feasibility and acceptability of delivering SBRT in this setting.

DETAILED DESCRIPTION:
Oligometastases or oligoprogression of ovarian cancer while on a PARPi may occur due to a secondary sub-clonal mutation causing acquired resistance in a small volume of tumour rather than having global tumour resistance. Eradication of the resistant disease with stereotactic radiotherapy (SBRT) would enable continuation of the PARPi to maintain control of disease that has retained drug sensitivity and this has the potential to impact disease outcomes.

For the purposes of this ovarian cancer trial, oligoprogression refers to the situation whereby 3 or less lesions of disease show evidence of progression. If there were previously other sites of disease, these remain in response or stable. Oligometastatic disease refers to the situation whereby complete response to treatment has been obtained and the disease relapse occurs that is limited in number and distribution (≤3 metastatic/recurrent lesions).

SOPRANO will explore whether there is activity of SBRT and SBRT followed by niraparib in the case of oligometastatic or oligoprogression disease post prior PARPi in recurrent ovarian cancer.

The trial will recruit patients with oligometastic or oligoprogressive ovarian cancer (≤3 sites/lesions) who have progressed on or following at least 6 months of treatment with PARP Inhibitor (PARPi). Patients will be randomised to one of two parallel non-comparative treatment cohorts:

* Cohort 1: SBRT followed by niraparib
* Cohort 2: SBRT alone

In both cohorts, therapy will continue until disease progression deemed by the investigator to warrant a change in treatment, unacceptable toxicity, withdrawal of consent or if the investigator decides it is not in the best interest of the patient to continue.

Adverse events, including toxicity from trial treatment will be collected and graded according to The National Cancer Institute (NCI) Common Terminology Criteria (CTC) Version 5.0 (http://ctep.cancer.gov/reporting/ctc.html).

Participants will be asked to consent for future linkage with routinely collected health data via national registries to trace their eventual vital status and assess subsequent unexpected comorbidities.

Assessment of disease by RECIST will be required 8 weekly following completion of SBRT for the first year and 12 weekly thereafter until disease progression meeting the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age.
2. Histologically confirmed epithelial ovarian, fallopian tube or primary peritoneal cancer.
3. Radiological disease progression whilst on, or following, any prior PARP inhibitor therapy. The PARP inhibitor is required to have been the patient's last systemic therapy.
4. Minimum duration of 6 months PARP inhibitor therapy as first line therapy or treatment for recurrent disease.
5. ≤3 lesions of progressive disease.
6. Each lesion to undergo SBRT <4 cm axial diameter, and feasible for SBRT as discussed in the SOPRANO virtual MDT (vMDT) meeting.
7. Measurable disease by RECIST criteria v1.1, which can be accurately assessed at baseline by CT or MRI. Patients with CA125 progression in the absence of measurable disease will NOT be eligible.
8. No contra-indication to restarting a PARP inhibitor.
9. Patients for whom surgery for recurrent disease is not planned.
10. Adequate baseline organ function to allow SBRT to all relevant targets as deemed by the investigator.
11. ECOG performance status of 0 or 1.
12. Predicted life expectancy ≥ 6 months.
13. Women of child-bearing potential who are confirmed NOT to be pregnant. This should be evidenced by a negative urine or serum pregnancy test within 72 hours prior to start of trial treatment. Patients will be considered to be not of child-bearing potential if they are:

    1. Post-menopausal -- defined as aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments, OR women under 50 years old who have been amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments and have serum follicle- stimulating hormone (FSH), luteinizing hormone (LH) and plasma oestradiol levels in the post-menopausal range for the institution.
    2. Able to provide documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.
    3. Radiation or chemotherapy-induced oophorectomy or menopause with > 1 year since last menses.
14. Willingness to commit to scheduled visits, treatments plans, laboratory tests and trial procedures.
15. Histological tissue specimen (tissue block or 8-10 unstained slides) must be available prior to commencing SBRT (specimen can be the sample at diagnosis or taken at relapse or progression). Otherwise, a biopsy must be carried out to obtain sufficient tissue for translational analyses.
16. Able to swallow, absorb and retain oral medication.
17. Able to provide written, informed consent.

Exclusion Criteria:

1. Co-morbidities which would preclude the safe use of SBRT.
2. Progressing or newly diagnosed brain metastases identified at the time of trial entry, not amenable to radical surgery or stereotactic radiosurgery. Previously treated brain metastases (i.e. palliative radiotherapy or systemic therapy) which have remained clinically and radiologically stable for ≥ 6 months are permissible.
3. Prior radiotherapy near the oligometastatic / oligoprogressive lesion precluding ablative SBRT. Suitability of lesions for ablative SBRT as part of the trial defined in Section 6.1 of this document and will be determined by the SOPRANO virtual MDT.
4. Treatment with any other investigational medicinal product (IMP) within the 4 weeks prior to trial entry.
5. Pregnant or lactating women.
6. Women of childbearing age and potential who are not willing to use a highly effective contraceptive measure.
7. Any unresolved toxicities from prior therapy should be no greater than CTCAE Grade 1 with the exception of Grade 2 alopecia or chemo-induced neuropathy at trial entry.
8. Clinical/radiological evidence of bowel obstruction (e.g. hospitalisation) or symptoms of sub-acute bowel obstruction within 6 weeks prior to trial entry.
9. Any other malignancy which has been active or treated within the past 3 years, with the exception of non-melanoma skin cancer. If prior treatment for another malignancy has taken place, then confirmation of ovarian/fallopian tube/peritoneal cancer progression is required e.g. biopsy, and discussion with the trial Chief Investigator and SBRT Lead
10. Judgment by the Investigator that the patient is unsuitable to participate in the trial and/or the patient is unlikely to comply with trial procedures, restrictions and requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 42 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | The primary timepoint of most interest for PFS is at six months after randomisation
  Progression free survival is defined as time from randomisation to evidence of progression of cancer at any site or death from any cause. Progression events should be imaging defined in all tumour types according to RECIST v1.1 criteria. Where SBRT specific consensus response assessment criteria exist for specific sites (e.g. spine), progression of SBRT treated lesions will be defined according to these guidelines.

SECONDARY OUTCOMES:
Time to first subsequent systemic therapy | Time to first subsequent systemic therapy assessed up to 2 years after randomisation.
  Time to first subsequent systemic therapy is defined as time from randomisation to commencing next systemic line of therapy or death from any cause (if this occurs before commencement of first subsequent treatment).
Time to first subsequent anti-cancer therapy | Time to first subsequent anti-cancer therapy assessed up to 2 years after randomisation.
  Time to first subsequent anti-cancer therapy is defined as time from randomisation to commencing next line of therapy (local or systemic) or death from any cause (if this occurs before commencement of first subsequent treatment).
Overall survival | The primary timepoint of interest for OS is at two years after randomisation.
  Overall survival (OS) defined as time from randomisation to death from any cause.
Local control at site of SBRT | Local control at site of SBRT assessed up to 2 years after randomisation.
  Local control at site of SBRT is defined as time from randomisation until radiological evidence of progression at the treated site and be measured on a lesion based analysis using RECIST v1.1 criteria
Time to 'Out of SBRT field' progression | Time to 'Out of SBRT field' progression assessed up to 2 years after randomisation.
  Time to 'Out of SBRT field' progression is defined as time from randomisation until radiological evidence of progression outside of treated area(s) for SBRT treatment using RECIST v1.1.
Clinician reported acute and late toxicity | Acute events are defined as those occurring up to 3 months follow up; late events are reported from 6 months post randomisation.
  Clinician reported acute and late toxicity will be graded using NCI CTCAE v5.0. Adverse events will be collected from start of treatment to disease progression (and 30 days post last dose of Niraparib for patients in cohort 1.
Quality of Life Assessments - FACT-O | Quality of Life will be collected at baseline prior to start of SBRT treatment, 4 weeks post SBRT treatment, 16, 24 and 48 weeks post randomisation and at disease progression.
  Functional Assessment of Cancer Therapy - Ovarian (FACT-O): FACT-O is a self-report measure that assesses physical well-being, social/family well-being, emotional well-being, functional well-being and ovarian cancer-specific subscale. The higher the score, the better the QOL.
  Quality of Life will be collected at baseline prior to start of SBRT treatment, 4 weeks post SBRT treatment, 16, 24 and 48 weeks post randomisation and at disease progression. Changes from baseline at each time point will be compared within groups as well as between treatment cohorts.
Quality of Life Assessments - EQ5D | Quality of Life will be collected at baseline prior to start of SBRT treatment, 4 weeks post SBRT treatment, 16, 24 and 48 weeks post randomisation and at disease progression.
  EQ-5D-5L: The EQ-5D-5L is a self-assessed, health related, quality of life questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The higher the score, the better the QOL.
  Quality of Life will be collected at baseline prior to start of SBRT treatment, 4 weeks post SBRT treatment, 16, 24 and 48 weeks post randomisation and at disease progression. Changes from baseline at each time point will be compared within groups as well as between treatment cohorts.
Feasibility of recruitment rate for the trial | Recruitment is expected to be over 2.5 years
  Feasibility of recruitment is defined as the recruitment rate for the trial
Proportion of patients receiving SBRT in the absence of new developing widespread disease | Proportion of patients receiving SBRT in the absence of new developing widespread disease assessed up to 2 years after randomisation.
  Proportion of patients receiving SBRT in the absence of new developing widespread disease, defined as greater than or equal to 4 metastatic sites, regional or distant, or a combination thereof.

OTHER OUTCOMES:
Time to widespread metastatic disease | Time to widespread metastatic disease assessed up to 2 years after randomisation.
  Time to widespread metastatic disease will be measured from the time of randomisation until radiological evidence of widespread metastatic disease, defined as greater than or equal to 4 metastatic sites, regional or distant, or a combination thereof.
Time to second subsequent therapy | Time to second subsequent therapy assessed up to 2 years after randomisation.
  Time to second subsequent therapy is defined as time from initiation of first subsequent therapy to commencing second line of therapy (local or systemic) or death (if this occurs before commencement of second subsequent treatment).
Mechanisms of PARP inhibitor resistance, immune-mediated effects, radiosensitivity and toxicities | From date of randomisation until date of progression meeting the primary endpoint or date of death from any cause, whichever came first, assessed up to 2 years
  Measurement of potential mechanisms of PARP inhibitor resistance, immune-mediated effects, radiosensitivity and toxicities. Measured between baseline and 4 weeks post-SBRT, 16, 24 and 48 weeks post randomisation, and disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Susana Banerjee, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (5):
- United Kingdom (5):
  - Western General Hospital, Edinburgh, Scotland
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - University College London Hospitals, London, UK
  - The Royal Marsden NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No